CLINICAL TRIAL: NCT05707650
Title: Reverse Breech Extraction Versus Push Technique for Fetal Delivery When Fetal Head is Deeply Impacted in the Pelvis During CS on A Fully Dilated Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ebtihal Ahmed, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS492/2021
Record Dates: First submitted 2023-01-15; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Obstructed Labor at Second Stage of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women allocated to this group will deliver by using reverse breech extraction technique. (Active Comparator)
  Interventions: Procedure: reverse breech extraction technique or push technique
- Women allocated to this group will deliver by using Push technique. (Active Comparator)
  Interventions: Procedure: reverse breech extraction technique or push technique

INTERVENTIONS:
Procedure: reverse breech extraction technique or push technique — using reverse breech extraction technique or push technique for disimpaction of fetal head during cs of a fully dilated cervix

SUMMARY:
Management of impacted fetal head during second stage cesarean requires careful and gentle attention to various surgical steps for delivery of a fetus without adverse maternal and neonatal outcomes, mostly by an experienced surgeon as in such situations, the lower uterine segment may be over-distended and indistinguishable from the vagina. Therefore, the uterine incision may inadvertently be placed too low, or in the vagina.

Also, it may be difficult for the operating surgeon to maneuver his hand below the deeply engaged fetal head, which may be further compounded by the presence of molding and edema on the fetal head (caput succedaneum).

This prospective controlled study was conducted at labor ward of department of obstetrics and gynecology at Ain Shams University Maternity Hospital to compare between the two techniques. A total of 70 pregnant women were enrolled and divided into two equal groups.

ELIGIBILITY:
Inclusion Criteria:

* • Singleton pregnancies.

  * Cephalic presentation will undergo cesarean section in advanced labor with the fetal head deeply engaged in the pelvis defined as fully dilated cervix and vertex at or below zero station

Exclusion Criteria:

* • Twins Pregnancies.

  * Breech or transverse presentation.
  * Woman has other obstetric indication to cs ex, fetal distress.
  * Woman has risk factor for bleeding ex, bleeding disorders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Uterine incision extension | intra-operative
  uterine extensions will include angle extensions on lower segments and into the broad ligaments".

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medecine At Ain Shams University, Cairo, Egypt